CLINICAL TRIAL: NCT05399667
Title: Assessment of Body Composition in Premature Children Submitted to an Early Stimulation Program
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0809
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Preterm Birth; Very Low Birth Weight Infant; Early Intervention; Parent-Child Relations; Nutrition, Healthy
Keywords: prematurity; very low birth weight; early intervention; parent-child relations; nutritional health; body composition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Early stimulation: Skin-to skin care by mother, kangaroo care, breastfeeding policy plus massage therapy are made by the mothers until hospital discharge. After discharge, they receive standard follow up care plus orientation for a continuous global simulation at home (total of 10 home visits independently of the standard evaluation and care that will be performed; visits promoting guidance and supervision sessions).
  Interventions: Other: Early stimulation
- Conventional care: Standard care according to the routine care of the Neonatal Intensive Care Unit (NICU) (skin-to skin care by mother, kangaroo care, and breast feeding policy) and their needs in the follow up program (motor, and cognition evaluations and interventions).
  Interventions: Other: Conventional care
- Control group: Term born children to obtain reference values for the variables evaluated in the present study.

INTERVENTIONS:
Other: Early stimulation — Preterm born children submitted to skin-to skin care (kangaroo care ) plus massage therapy by their mothers. This group received tactile-kinesthetic stimulation by mothers from randomization until hospital discharge. Intervention performed exclusively by the mothers was based on studies regarding the application of skin stimulations and passive exercises in preterm infants
  Groups: Early stimulation
Other: Conventional care — Preterm born children submitted to skin-to skin care by their mothers (kangaroo care), associated to standard care according to the routine care in the Neonatal Intensive Care Unit (NICU).
  Groups: Conventional care

SUMMARY:
This is a cross-sectional study of a randomized clinical trial to investigate nutritional aspects of pre-scholar aged children born preterm submitted to an early stimulation program versus conventional care program. The preterm-born children participated in the project entitle "Early Intervention Program for Preterm Infants and Their Parents: establishing the impact at 18 Months Corrected Age" (NCT02835612), which performed a continuous early stimulation in very and extremely preterm infant's families in their first 12 to 18 months. In the present study, preterm born children currently with 3 to 6 years old and their mothers (or legal guardian) are once more invited to a one-day visit for a nutritional and clinical evaluation at the Clinical Research Center of Hospital de Clínicas de Porto Alegre/Brazil. In the consultation, preterm born children and theirs mothers are submitted to the following exams: body composition by electrical bioimpedance, clinical and physical evaluation, anthropometric measurements, and children's eating habits, eating behavior and parental educational style in food through specific questionnaires. Moreover, this study will also investigate a group of pre-scholar health children born at term to obtain reference values for variables analysed. The goal with these findings is to determine if an early stimulation program could present a positive impact in anthropometric outcomes and nutritional aspects in this more vulnerable preterm born population.

DETAILED DESCRIPTION:
The main goal of the present study is to investigate anthropometric and physical measurements of pre-scholar aged children born preterm and their parents submitted to an early stimulation program, as well as to investigate children's eating practices, children's eating behavior and parental educational style in feeding.

This currently study is a segment of a previous project entitle: Early Intervention Program for Preterm Infants and Their Parents: establishing the impact at 18 Months Corrected Age (NCT02835612), which performed a continuous early stimulation in very preterm infant's families in their first 12 to 18 months. The previous study randomized preterm born children less than 32 weeks of gestational age and/or very low birth weight at Hospital de Clínicas de Porto Alegre (HCPA) - a tertiary hospital in south Brazil, in the following two groups: CONVENTIONAL GROUP (CG) that received standard care (skin-to skin care by mother, kangaroo care, and breast feeding policy) according to the routine care of the Neonatal Intensive Care Unit (NICU) and, after NICU discharge, they were referred for a traditional follow up clinic taking care of the demands according to their necessity. INTERVENTION GROUP (IG): Skin-to skin care by mother, kangaroo care, breastfeeding policy plus massage therapy were made by the mothers until hospital discharge. After discharge, they received standard follow up care plus orientation for a continuous global simulation at home. The early intervention was performed according to developmental milestones, anticipating in one month evolutional step acquisition of motor and/or cognitive expected for corrected age. Besides that, we have a total of 10 home visits promoting guidance and supervision sessions.

In the present study, preterm born children aging between 3 to 6 years old and their mothers (or legal guardian) are once more invited to a one-day visit in the Clinical Research Center of HCPA for nutritional and clinical evaluation. In the visiting day, research participants are submitted to the following exams: body composition by electrical bioimpedance (InBody 770), anthropometric measurements (weight, height, skinfold thickness), clinical and physical evaluation (6 minutes walt test) and children's eating habits, eating behavior and parental educational style in food through specific questionnaires, such as Behavioral Pediatrics Feeding Assessment Scale (BPFAS), Child Eating Behaviour Questionnaire (CEBQ) and Caregiver's Feeding Styles Questionnaire (CFSQ). Data from neonatal period and from the follow up in the clinical care will also be analysed to associate with current nutritional and clinical findings. In addition to preterm population, a group of term born health children and their mother will be invited to participate with the goal to access reference values of the parameters investigated. This group of term born children (>37 weeks of gestational age and/or birth weight >2500g) will be recruited from the daycare of our hospital institution.

It is expect with these findings to determine if an early stimulation program could present a positive impact in anthropometric outcomes and nutritional aspects of our more vulnerable preterm born population.

ELIGIBILITY:
Inclusion Criteria: Preterm children born at HCPA (birth weight <1500g and/or gestational age <32 weeks); Term born children (> 37 weeks of gestational age and/or birth weight >2500g)

Exclusion Criteria: Congenital malformations

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm born children aging 3 to 6 years old who were born at Hospital de Clínicas de Porto Alegre and their mother.
  Term born children aging 3 to 6 years old who are in the Daycare for the employes of the Hospital de Clínicas de Porto Alegre.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Body composition | 1 day of evaluation
  Body composition is evaluated by bioelectrical impedance analysis (BIA) (InBody 770, Biospace Co Ltd). Each participant is positioned in an orthostatic position on a platform with lower electrodes for the feet and the hands holding onto upper electrodes. The measurement is performed after 2 hours fasting and diapers are changed before the evaluation.

SECONDARY OUTCOMES:
Child Eating Behaviour | 1 day of evaluation
  Children's eating behavior is evaluated with the Brazilian validated and translated Children's Eating Behavior Questionnaire (CEBQ). The CEBQ is a Likert-type, parent-report rating scale measuring the variation in eating behavior in children, and consists of 35 items comprising eight subscales (Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating, and Food fussiness). Parents are asked to rate their child's eating behavior on a five-point scale (never, rarely, sometimes, often, always; 1-5, respectively). A higher mean score for each specific sub-scale suggests the child shows a higher tendency toward the respective eating behavior.
Individual differences in parenting feeding styles | 1 day of evaluation
  Parents should complete the 19-item Child Feeding Styles and Practices Questionnaire (CFSQ). Each item is scored from 1 (never) to 5 (always). Scores are averaged and categorized into one of four feeding styles: authoritative, authoritarian, indulgent, and uninvolved; higher scores represent more of the feeding style.
Nutritional Assessment in Behavioral Pediatrics | 1 day of evaluation
  Behavioral Pediatrics Feeding Assessment Scale (BPFAS) is a parent-report questionnaire with 35 questions, which examines the frequency of child behaviors (e.g., will try new foods) and frequency of parent feelings and strategies for dealing with eating problems (e.g., frustration when feeding a child, cajoling or threatening in response to frustration when feeding) using a five-point Likert scale from "never" to "always." Parents are also asked to rate whether each item is a problem by answering with a "yes" or "no".
Feeding practice | 1 day
  The child's eating habits are evaluated through a questionnaire that seeks to understand the quality of food since birth. This questionnaire comprises information on breastfeeding, use of infant formula, and food introduction, including the period when 20 specific foods were introduced. They are sugary foods, treats, protein sources, caffeine, and vegetables. In addition to this questionnaire, a 24-hour food recall of the child is requested.
Anthropometric evaluation of children and a parent respecting body weight. | 1 day of evaluation
  The trained research team measures the body weights (in kilograms = kg) of the children and a parent with the method described by the World Health Organization (WHO) using the same measuring instruments. Measurements are performed using a standardized digital scale U.R. 10.000 Light.
Anthropometric evaluation of children and a parent respecting height. | 1 day of evaluation
  The trained research team measures the height (in centimeters = cm) of the children and a parent, using the same wall stadiometer Sanny®, with individuals in an upright position, their heels, back, and head touching the equipment, the latter in a Frankfort plane.
Anthropometric evaluation of children and a parent respecting skinfold. | 1 day of evaluation
  The trained research team measures the skinfolds of the children and a parent, measured with a skinfold caliper Lange®, using the anthropometry technique described by ISAK. The subscapular and triceps skinfolds are measured.
Anthropometric evaluation of children and a parent respecting circumferences. | 1 day of evaluation
  The trained research team measures the circumferences of the children and a parent using a measuring tape. Waist and arm circumference is evaluated in all individuals, as well as head circumference in children.
Z-score calculations of all participants using WHO ANTHRO program. | 1 day of evaluation
  The anthropometric (height-for-age, weight-for-age; body mass index-for-age) measurements are evaluated according to the Z-score using the WHO ANTHRO program and WHO ANTHRO Plus Software.
Physical Activity questionnaire | 1 day of evaluation
  The questionnaire estimates the sedentary and active time of children, separated into weekdays or weekends, and day shifts (morning, afternoon, and night). The measure of physical activity is expressed by the daily time of participation in games and outdoor play while the measure of sedentary behavior is based on the time of watching television.
Physical capacity Assessment | 1 day of evaluation
  Physical capacity using Six Minutes Walk Test following the guidelines of American Thoracic Society (ATS), in a corridor of 30 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana R Bernardi, Prof PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrews ET, Beattie RM, Johnson MJ. Measuring body composition in the preterm infant: Evidence base and practicalities. Clin Nutr. 2019 Dec;38(6):2521-2530. doi: 10.1016/j.clnu.2018.12.033. Epub 2019 Jan 12. PMID 30737045
- [Background] Hughes SO, Cross MB, Hennessy E, Tovar A, Economos CD, Power TG. Caregiver's Feeding Styles Questionnaire. Establishing cutoff points. Appetite. 2012 Feb;58(1):393-5. doi: 10.1016/j.appet.2011.11.011. Epub 2011 Nov 15. PMID 22119478
- [Background] Saenz de Pipaon M, Dorronsoro I, Alvarez-Cuervo L, Butte NF, Madero R, Barrios V, Coya J, Martinez-Biarge M, Martos-Moreno GA, Fewtrell MS, Argente J, Quero J. The impact of intrauterine and extrauterine weight gain in premature infants on later body composition. Pediatr Res. 2017 Oct;82(4):658-664. doi: 10.1038/pr.2017.123. Epub 2017 Jul 5. PMID 28678222
- [Background] Crist W, Napier-Phillips A. Mealtime behaviors of young children: a comparison of normative and clinical data. J Dev Behav Pediatr. 2001 Oct;22(5):279-86. doi: 10.1097/00004703-200110000-00001. PMID 11718230
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Silveira RC, Mendes EW, Fuentefria RN, Valentini NC, Procianoy RS. Early intervention program for very low birth weight preterm infants and their parents: a study protocol. BMC Pediatr. 2018 Aug 9;18(1):268. doi: 10.1186/s12887-018-1240-6. PMID 30092772
- [Background] Oliveira NKR de, Lima RA de, Mélo EN, Santos CM, Barros SSH, Barros MVG de. Reliability of a questionnaire to assess physical activity and sedentary behavior in preschool-aged children. Rev. Bras. Ativ. Fís. Saúde [Internet];2011; 16(3):228-33. https://rbafs.org.br/RBAFS/article/view/597